CLINICAL TRIAL: NCT04724564
Title: Correlation of Different Time Measurements of the Surgical PLETH Index With Postoperative Pain; a Prospective Observational Study
Brief Title: Correlation of Different Time Measurements of the Surgical PLETH Index With Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate Professor of Anesthesiology, Fayoum University Hospital
Other Study IDs: M 703
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Abdominal Hysterectomy
Keywords: Hysterectomy; Analgesic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: THE SURGICAL PLETH INDEX — CORRELATION OF DIFFERENT TIME MEASUREMENTS OF THE SURGICAL PLETH INDEX WITH POSTOPERATIVE PAIN

SUMMARY:
Despite the major progress in anesthetic techniques, postoperative pain is still considered a major problem during practice. (1-3). Leading to many co-morbidities, one to two-thirds of patients will suffer postoperative pain. These co-morbidities can include; pulmonary complications, cardiac complications, and delirium(4). Numerous risk factors are associated with the emergence of postoperative pain, including; younger age, female sex, preoperative pain, and extensive surgical procedure. The severity of postoperative pain may vary among patients undergoing the same operation (5-10).

Many techniques have been evolved to monitor nociception and predict postoperative pain intensity; one of the most recent techniques is the surgical pleth index (SPI)(11).SPI is a noninvasive dimensionless score; its value is obtained from heartbeat interval and pulse wave amplitude monitored by pulse oximetry probe.SPI reflects the sympathetic response of the patient to the surgical stimuli(12-13). It was reported that SPI is better than other parameters like heart rate and blood pressure for detecting the balance between nociceptor activation and analgesia(14-15), and its value is correlated with the severity of postoperative pain. SPI values range from 0 to 100, and higher values indicate strong surgical stimulus (16). SPI can be used as a guide for intraoperative analgesia; hence, it can be a valuable tool to assess the analgesic requirement and limit opioid consumption, both preoperative and postoperative(17).

Several studies have been performed to predict the severity of postoperative pain using SPI in adults and children (16,18). It was also used successfully to expect a hemodynamic response to tracheal intubation and skin incision (19) and monitor nerve block success. (20).

However, since SPI has emerged, the most sensitive cut-off value that correlates well with postoperative pain severity remained debatable. Recent studies reported a value of 30 as a cut-off value of SPI. (21). On the other hand, the time of measurement to rely on was debatable. Most studies recommended that a measure of SPI before recovery can be used. However, a more recent study suggested that SPI response to surgical incision is highly correlated with postoperative pain and opioid consumption (18). Based on these data, we hypothesized that both measurements are correlated with postoperative pain and aimed to test which measure is more correlated.

DETAILED DESCRIPTION:
The current study's objective is to determine the optimum time to measure intraoperative SPI, which correlates better with postoperative pain.

Methods:

The study will be performed at Fayoum university hospital after the local institutional ethics committee and local institutional review board's approval. The study design will be a prospective observational study.A total of 99 patients scheduled for elective abdominal hysterectomy under general anesthesia and their age range from 18-65 will be included in this trial.

Exclusion criteria included; an age <18 years, significant dysrhythmia like AF or atrioventricular block more than1st degree, patient with a pacemaker,treatment with vasoactive medications, and any intraoperative t reatment with clonidine, beta-receptor agonists or antagonists, or anyother drug that can affect the sympathovagal balance.patients receiving neuraxial anesthesia will also be excluded.

Anesthesia and pain management:

All patients will fast 6 hours for solid food and 2 hours for clear fluids before the operation. After arriving the operating room, standard monitoring (Pulse oximetry, Noninvasive blood pressure, and Electrocardiogram)will be applied and continued all over the operation. An 18G peripheral cannula will be inserted.All patients will be pre-oxygenated with 100% O2 and premedicated with 0.03 mg/kg IV midazolam and10 mg metoclopramide. Intravenous induction of anesthesia will be performed using2mg/kg propofol, l-2µgm/kg fentanyl and0.5mg/kg atracurium. All patients will receive 1gm paracetamol IV as intraoperative supplementary analgesia just after the induction. An endotracheal tube will be inserted for all patients. Mechanical ventilation will be adjusted as volume controlled ventilation with 5cmH2oaiming to maintain end-tidalCo2 pressure of 30 to 40 mmHg by a mixture of O2with fiO20.5and air. Anesthesia will be maintained with isoflurane. SPI will be recorded 5 min after skin incision and 10 min before recovery. Using anesthesia machine( carestatation 650 l GE.3.4.2019) After recovery,Upon ability of communication, all patients will be asked to quantify their level of pain on a 0 - 10 point numeric rating scale (NRS) with (0= no pain, 1-3 mild, 4-5 moderate and 6-10 severe) three scores will be obtained with 5 minutes intervals and the highest pain score of the three will be recorded for further analysis (without affection of the routine pain management).

All patients will be transferred to the obstetrics ward when they reach a modified Aldrete score ≥9. During the first 24 hours, all patients will receive IV paracetamol 1 g every 8 hours for postoperative analgesia according to the obstetric department protocol. In addition to intravenous tramadol through PCA

(concentration of 4 mg/ml) with 20 mg dose, 10 minutes lockout interval, and one hour limit of 50 mg.

Measured parameters:

SPI at 5 minutes after skin incision and 10 minutes before recovery, the highest pain score (NRS) in the PACU,total opioid consumption during the first 24 hours, Nausea and vomiting (will be assessed on a scale: 0 = no symptoms, 1 = only nausea, 2 = nausea and/vomiting), Respiratory depression (will be defined as respiratory rate lower than 10), Sedation (will be assessed using a sedation score where 0 = awake and alert, 1 = quietly awake, 2 = asleep but easily arousable, 3=deep sleep, responding to a painful stimulus) All these data will be collected by a separate anesthesiologist who will be blinded with the study.

The primary outcome is to determine which SPI measurement is more correlated with postoperative pain. The secondary outcomes is to evaluate the correlation between the SPI measurements and opioid consumption in the first postoperative 24 hours and to define the cut-off value of SPI measurements

ELIGIBILITY:
Inclusion Criteria:

* elective abdominal hysterectomy under general anesthesia and their age range from 18-65

Exclusion Criteria:

* an age <18 years
* significant dysrhythmia like AF or atrioventricular block more than1st degree
* patient with a pacemaker
* treatment with vasoactive medications, and any intraoperative treatment with clonidine, beta-receptor agonists or antagonists, or any other drug that can affect the sympathovagal balance.
* Patients receiving neuraxial anesthesia

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-65 year
Study Population: patients admitted in Fayoum uniersity hospital who are candidates for elective abdominal hysterectomy under general anesthesia and their age range from 18-65
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
which SPI measurement is more correlated with postoperative pain | SPI at 5 minutes after skin incision and 10 minutes before recovery
  The primary outcome is to determine which SPI measurement is more correlated with postoperative pain

SECONDARY OUTCOMES:
the correlation between the SPI measurements and opioid consumption | the first postoperative 24 hours
  the correlation between the SPI measurements and opioid consumption
the cut-off value of SPI measurements | SPI at 5 minutes after skin incision and 10 minutes before recovery
  to define the cut-off value of SPI measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Fayoum University Hospital
Locations (1):
- Fayoum University hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
No plane to share IPD

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Persson AK, Dyrehag LE, Akeson J. Prediction of Postoperative Pain From Electrical Pain Thresholds After Laparoscopic Cholecystectomy. Clin J Pain. 2017 Feb;33(2):126-131. doi: 10.1097/AJP.0000000000000394. PMID 27258997
- [Background] Persson AKM, Akeson J. Prediction of Acute Postoperative Pain from Assessment of Pain Associated With Venous Cannulation. Pain Pract. 2019 Feb;19(2):158-167. doi: 10.1111/papr.12729. Epub 2018 Nov 5. PMID 30269418
- [Background] Jung K, Park MH, Kim DK, Kim BJ. Prediction of Postoperative Pain and Opioid Consumption Using Intraoperative Surgical Pleth Index After Surgical Incision: An Observational Study. J Pain Res. 2020 Nov 6;13:2815-2824. doi: 10.2147/JPR.S264101. eCollection 2020. PMID 33192089